CLINICAL TRIAL: NCT07097779
Title: A Comparison of Visual Aids for Stroke Rehabilitation: Photos, Videos, Pictograms
Brief Title: Helping Stroke Patients With Movement Using Photos, Videos, and Pictograms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaegyeong Lee (Other)
Responsible Party: Sponsor-Investigator, Jaegyeong Lee, Principal Investigator, Sahmyook University
Organization: Sahmyook University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYU 2025-06-028-003
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Stroke
Keywords: Pictograms; Cognitive load; Visual aids; Motor performance; Photos; Videos; Visual instruction; Movement accuracy
MeSH Terms: conditions — Stroke | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Visual Aids Intervention (Experimental)
  Interventions: Behavioral: Visual Aids(Photos, Videos, and Pictograms)

INTERVENTIONS:
Behavioral: Visual Aids(Photos, Videos, and Pictograms) — Participants will be presented with three types of visual instructional aids: photographs, videos, and pictograms, via a laptop or tablet. Each participant will perform three motor tasks, each paired with a different visual aid, assigned in random order using a Latin Square design. Each task takes approximately 3 minutes, followed by 1 minute of rest. After completing all tasks, participants will complete a 5-minute survey about their understanding, preference, and perceived cognitive load. The total session lasts about 20 minutes.

SUMMARY:
The goal of this interventional study is to learn how different types of visual aids-photos, videos, and pictograms-help people with stroke understand and perform simple physical movements. The researcher wants to find out which type of visual aid is most helpful and easiest to understand for stroke rehabilitation.

To take part, participants must be able to stand for at least one minute without help and understand simple instructions.

The main questions this study aims to answer are:

* Which type of visual aid (photo, video, or pictogram) helps participants perform movements more accurately?
* Which visual aid do participants find the easiest to understand and prefer?
* How much mental effort (cognitive load) do participants feel when using each type of visual aid?
* Do the effects of visual aids vary depending on stroke type, brain lesion location, or time since stroke?

The researcher will compare how each type of visual aid affects movement performance and participants' responses.

Participants will:

* View three types of visual aids (photo, video, pictogram) and perform specific physical tasks based on each.
* Have their movement performance recorded using a video camera.
* Complete a short survey after the tasks to rate their understanding, preferences, and cognitive effort.
* Take part in a single session that lasts about 20 minutes in a quiet room within the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stroke.
* Have sufficient vision and cognitive ability to perceive the provided visual materials (pictures or text).
* Able to stand independently without assistive devices for at least 1 minute.
* Have minimum cognitive ability necessary to understand tasks and follow instructions, with a score of 18 or higher on the Korean version of the Mini-Mental State Examination (K-MMSE).

Exclusion Criteria:

* ndividuals with other central nervous system disorders besides stroke that may affect motor performance or assessment.
* Individuals with musculoskeletal disorders, such as arthritis or fractures, that may affect motor performance or assessment.
* Individuals with severe visual impairments, such as visual field defects, unilateral neglect, or color blindness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-09-06 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-11-09 (Actual)

PRIMARY OUTCOMES:
Motor Task Performance Accuracy | Immediately after the experimental session
  Motor task performance accuracy will be assessed using a checklist developed by the researchers, considering task characteristics and learning effects. Each movement consists of 6 key performance elements, scored as 0 (not performed) or 1 (performed accurately), with a maximum of 6 points per task. All performances will be video recorded, and three trained raters will independently score the recordings. Inter-rater reliability will be evaluated using the Intraclass Correlation Coefficient (ICC) based on total scores.

SECONDARY OUTCOMES:
Number of Replays | During each task trial (approximately 3 minutes per task)
  The number of times the participant presses the replay button to review the visual instructional material before performing the task will be automatically recorded. This measure will be stored using PsychoPy 2025.1.1 (Open Science Tools Ltd., Nottingham, UK).
Number of Hesitations | Immediately after the experimental session (video review)
  The number of hesitations will be counted during motor task performance. A hesitation is defined as a pause lasting more than 1 second, re-checking the visual aid, or modifying the movement. This measure indirectly reflects the participant's movement fluency and level of cognitive certainty. All performances will be video recorded and independently reviewed by three trained raters. Inter-rater reliability will be assessed using the Intraclass Correlation Coefficient (ICC 3,k).
Understanding of Visual Aids | Immediately after the experimental session
  Participants will rate how helpful each type of visual aid (photo, video, pictogram) was for understanding the motor task. A 5-point Likert scale will be used, where 1 indicates "Not helpful at all" and 5 indicates "Very helpful." Participants will complete this rating immediately after completing each task.
Preference for Visual Aids | Immediately after the experimental session
  Participants will indicate which of the three visual instructional aids (photos, videos, pictograms) they found easiest to understand. This measure captures participants' relative preference for the visual materials after performing the motor tasks.
Perceived Cognitive Load | Immediately after the experimental session
  The degree of mental effort experienced by participants while performing the motor tasks with each type of visual instructional material will be assessed. A pictorial 9-point Likert scale will be used, where a score of 1 indicates "not difficult at all" and a score of 9 indicates "very difficult"

CONTACTS AND LOCATIONS:
Locations (1):
- Ilsan Central Rehabilitation Hospital, Goyang-si, South Korea